CLINICAL TRIAL: NCT00306969
Title: Phase I/II Study of Oral Bexarotene in Combination With Photopheresis for Treatment of Cutaneous T-Cell Lymphoma
Brief Title: Study of Oral Bexarotene in Combination With Photopheresis for Treatment of Cutaneous T-Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Ligand Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2001-391G
Record Dates: First submitted 2006-03-23; First posted 2006-03-27 (Estimated); Last update posted 2006-03-27 (Estimated); Status verified 2004-09

CONDITIONS: Cutaneous T-Cell Lymphoma
Keywords: mycosis fungoides, Sézary Syndrome
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — Bexarotene; Photopheresis

INTERVENTIONS:
Drug: bexarotene
Device: photopheresis

SUMMARY:
This is a pilot study of the safety and tolerability of photopheresis in combination with increasing doses of oral bexarotene in patients with cutaneous T-cell lymphoma.Our hypotheses are that the combination of bexarotene with photopheresis is safe and that bexarotene will enhance immune response in the setting of extracorporeal photopheresis in the treatment of cutaneous T-cell lymphoma (CTCL), resulting in a shorter time to clinical response.

DETAILED DESCRIPTION:
Photopheresis is FDA-approved as a device in the treatment of patients with cutaneous T-cell lymphoma. Using treatment schedules of once monthly treatment, with each treatment consisting of two consecutive days of photopheresis, initial response rates of 20-60% have been reported. However, in publications, for those who attained a complete response, median time to response was 11 months (range 5 to 14 months). Response has been shown to correlate with intact immune function in patients with normal CD8+ cell prior to therapy. The mechanism of activity of photopheresis in cutaneous T-cell lymphoma while not fully understood involves apoptosis of malignant tumor cells. Modifications in the original scheduling of photopheresis, with shorter cycles of 2 or 3 weeks, have met with success. Several centers have been using an accelerated delivery schedule of treatments, treating patients every 2 weeks.

Bexarotene was FDA approved for patients with CTCL. It is an RXR selective retinoid. Retinoids can serve as physiologic rather than cytotoxic drugs to arrest or reverse the process of carcinogenesis. There is a growing body of evidence that supports a role for retinoids in the induction of apoptosis. In the two, completed Phase II-III studies that formed the basis of approval (approved dose is 300mg/m2/day) of bexarotene capsules, 193 patients with previously treated CTCL were administered bexarotene capsules. Response rates were in the order of 50% for the 300mg/2/day, however, 79% of patients had hyperlipidemia.

This study will therefore primarily examine the safety and tolerability of using increasing doses of bexarotene in combination with photopheresis. As a secondary endpoint, we will attempt to establish whether bexarotene can upregulate the immune response and therefore potentially enhance the response rates to photopheresis in patients with CTCL.

Six cohorts of patients will be treated:

Dose level cohorts enrollment will be sequential with centralized dose assignment at Boston Medical Center

To establish safety, a 30 day pause will occur between cohorts. During the 30 day waiting period, additional patients will be able to enter the open cohort, provided that there is no grade 3 or 4 toxicity in the 3 patients already entered into the cohort. Once the 30 day period has ended, new patients will be able to enter the next cohort.

Cohort 1 (3 patients): Bexarotene will be given at the dose of 75mg po per day with food for 7 days prior to beginning photopheresis(Day -6 to 0, day 1 being the day when photopheresis begins on first day of cycle 1). Photopheresis will be performed on 2 consecutive days the first 2 days of each 21 day cycle. Bexarotene will be given concurrently with photopheresis for 4 cycles. The duration of the study is 3 months with premature discontinuation for toxicity at the discretion of the investigator, or progressive disease.

Cohort 2 (3 patients): Bexarotene will be given at the dose of 150 mg po per day with food for 7 days prior to beginning photopheresis (Day -6 to 0, day 1 being the day when photopheresis begins on first day of cycle 1). Photopheresis will be performed on 2 consecutive days the first 2 days of each 21 day cycle. Bexarotene will be given concurrently with photopheresis for 4 cycles. The duration of the study is 3 months with premature discontinuation for toxicity at the discretion of the investigator, or progressive disease.

Cohort 3 (3 patients): Bexarotene will be given at the dose of 225 mg po per day with food for 7 days prior to beginning photopheresis (Day -6 to 0, day 1 being the day when photopheresis begins on first day of cycle 1). Photopheresis will be performed on 2 consecutive days the first 2 days of each 21 day cycle. Bexarotene will be given concurrently with photopheresis for 4 cycles. The duration of the study is 3 months with premature discontinuation for toxicity at the discretion of the investigator, or progressive disease.

Cohort 4 (3 patients): Bexarotene will be given at the dose of 300 mg po per day with food for 7 days prior to beginning photopheresis (Day -6 to 0, day 1 being the day when photopheresis begins on first day of cycle 1). Photopheresis will be performed on 2 consecutive days the first 2 days of each 21 day cycle. Bexarotene will be given concurrently with photopheresis for 4 cycles. The duration of the study is 3 months with premature discontinuation for toxicity at the discretion of the investigator, or progressive disease.

Cohort 5 (3 patients): Bexarotene will be given at the dose of 375 mg po per day with food for 7 days prior to beginning photopheresis (Day -6 to 0, day 1 being the day when photopheresis begins on first day of cycle 1). Photopheresis will be performed on 2 consecutive days the first 2 days of each 21 day cycle. Bexarotene will be given concurrently with photopheresis for 4 cycles. The duration of the study is 3 months with premature discontinuation for toxicity at the discretion of the investigator, or progressive disease.

Cohort 6 (3 patients): Bexarotene will be given at the dose of 450 mg po per day with food for 7 days prior to beginning photopheresis (Day -6 to 0, day 1 being the day when photopheresis begins on first day of cycle 1). Photopheresis will be performed on 2 consecutive days the first 2 days of each 21 day cycle. Bexarotene will be given concurrently with photopheresis for 4 cycles. The duration of the study is 3 months with premature discontinuation for toxicity at the discretion of the investigator, or progressive disease.

Toxicity will be assessed using the National Cancer Institute common Toxicity Criteria at the beginning of each 21 day cycle. Assessments will be every 3 weeks and at the final follow-up visit.

All patients will undergo a skin biopsy from lesional skin prior to entry to confirm active disease. A portion of the biopsy will be used for immunohistochemical studies to identify populations of activated lymphocytes in the skin and to identify apoptotic markers (TUNNEL METHOD). A skin biopsy will be subsequently obtained after 7 days of bexarotene, and at the end of the study. A portion of each skin biopsy will be used for immunohistochemical studies to identify populations of activated lymphocytes in the skin (TGF-B and Fas on malignant T cells) and to identify apoptotic markers (TUNNEL method)

All patients will undergo baseline studies of immune function, including a FACS analysis of circulating lymphocyte populations to identify activation antigens on T-lymphocytes, as well as in vitro assays of T-cell function such as proliferation assays and cytokine production by cultured T-cells. These studies will be repeated after the second and fourth. For these assays, one green top tube will be drawn on day 1 before photopheresis and on day 2 at the completion of therapy. One serum tube (one red top) will be drawn on days 1 and 2 and serum will be stored at -20° until the assays are performed.

In summary, the following research skin biopsies and labs will be obtained:

Baseline (Day -6): one green top and one red top Baseline (Day -6): skin biopsy from lesional skin

Day 1 of cycle 1: skin biopsy from lesional skin

Cycles 2 and 4: Day 1: one green top and one red top Day 2 one green top and one red top

End of cycle 4: skin biopsy from lesional skin

In addition to the following evaluations, the BASELINE visit will include a history with patient demographic. At the baseline, tri-weekly, and final visits, the following information will be collected:

* Patient weight.
* Serum chemistries, including LDH, LFTS, albumin, uric acid, Ca, Phos, Mg, Cholesterol, Triglycerides, Thyroid function (T4, TSH)
* CBC differential, Sezary count if applicable
* ECOG score.
* Skin assessment (previously published weighted skin score) and a description of other symptoms attributed to CTCL, and at the final visit, an overall assessment
* Names and doses of all concomitant medications
* Quality of Life assessment (Skindex-29 and FACT-G)

The investigator will also evaluate patient's response by organ system involvement, with an overall assessment, as follows:

* Complete Response (CR): Resolution of all manifestations of CTCL lasting one month.
* Partial Response (PR): A 50% improvement of the sum total of all disease (CTCL) lasting one month.
* No Change (NC): Failure to meet criteria for either response or progressive disease.
* Progression: a 25% or more progression of existing disease or the appearance of any new disease (disease worsening).
* Flare: After an initial response (either CR or PR), an increase in the manifestation of CTCL requiring additional treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have biopsy-proven CTCL. Stages of CTCL IIA or greater are eligible.
2. Patients with stage IB, either resistant to 2 prior therapies, resistant to 1 prior therapy and intolerant to a second one, or intolerant to 2 prior therapies, will also be eligible.
3. Patients previously treated with photopheresis will be eligible
4. Patients previously treated with oral or topical bexarotene will be eligible -a 1 month wash out period will be required prior to entry into the study
5. Measurable or evaluable disease.
6. Median life expectancy at least three months
7. Females of child bearing potential must consent to the use of 2 forms of reliable contraceptives, one of which must be non-hormonal.
8. All patients must provide written informed consent.
9. Patients must have completed any prior treatment at least 2 weeks before enrollment.
10. No concomitant medications for CTCL, including no topical steroids
11. Chronic topical steroid use is allowed if patients require low dose steroids for palliation of pruritus, but topical steroid therapy cannot be initiated after enrollment.
12. No history of myocardial infarction within six months, no history of unstable angina or unstable blood pressure
13. No oral or topical retinoid therapy within 1 month of entry in the study.
14. No history of pancreatitis or pancreatic disease or surgery
15. Fasting serum triglyceride within normal limits or "normalized" prior to study entry with appropriate intervention such as the use of an antilipid agent.

    * Cholesterol < 239 mg/dl
    * Triglyceride < 250 mg/dl
16. Patients must have adequate renal, hepatic, cardiac function and hematologic values:

    * CBC :WBC>2000, HGB>9, Plt >30K.
    * Chemistry panel: Creatinine <2.5, LFTS <3x NL, albumin>2.5.
    * Absence of hepatic dysfunction characterized by SGOT (AST), SGPT (ALT), or serum bilirubin >3 times the upper limit of normal
17. Women of child-bearing potential must have negative pregnancy test (serum *-HCG) with a sensitivity of at least 50 mIU within seven (7) days prior to the initiation of treatment and must have used effective contraception (recommended to be two reliable forms of contraception used simultaneously, at least one of which should be non-hormonal) or must have been sexually abstinent for at least four (4) weeks prior to the negative pregnancy test through entry in the study.

Exclusion Criteria:

The following patients are excluded:

* inability to safely tolerate temporary removal of up to 750 ml of circulating blood due to poor vascular disease or labile blood pressure
* pregnant, intent to become pregnant, or lactating females.
* known hypersensitivity to bexarotene or other component of bexarotene capsules.
* Risk factor for pancreatitis (e.g., prior pancreatitis, uncontrolled hyperlipidemia, excessive alcohol consumption, uncontrolled diabetes mellitus, biliary tract disease, and medications known to increase triglyceride levels or to be associated with pancreatic toxicity)
* No systemic vitamin A in doses exceeding 15,000 IU/day within 14 days prior to initiating bexarotene
* drug dependence or a psychiatric condition, which in the opinion of the investigator will interfere with participating in the study.
* ECOG performance status of 3 or greater.
* patients with known photosensitive disease.
* allergy to psoralen.
* patients with active uncontrolled infection.
* patients currently participating in another investigational study.
* patients with a systolic blood pressure £ 90 mmHg.
* Patients who do not meet eligibility criteria for laboratory studies
* Unwillingness or inability to minimize exposure to sunlight and artificial ultraviolet light while receiving bexarotene
* Unwillingness to agree to sexual abstinence or to comply with effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2001-12; Study Completion 2004-04

PRIMARY OUTCOMES:
Safety and tolerability of bexarotene in combination with ECP, assessed with NCI toxicity assessment, at each treatment visit, every 3 weeks and at final one month foll

SECONDARY OUTCOMES:
Time to response of bexarotene with ECP in patients with CTCL, at month 4 (follow-up visit) patient's response by organ system involvement, with an overall assessment: complete response, partial response, no change, or progressive disease, flare.
Another secondary outcome is whether combination of instruments provides relevant information on CTCL patients' health related quality of life during therapy

CONTACTS AND LOCATIONS:
Overall Officials: Marie-France Demierre, MD, Principal Investigator — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Duvic M, Martin AG, Kim Y, Olsen E, Wood GS, Crowley CA, Yocum RC; Worldwide Bexarotene Study Group. Phase 2 and 3 clinical trial of oral bexarotene (Targretin capsules) for the treatment of refractory or persistent early-stage cutaneous T-cell lymphoma. Arch Dermatol. 2001 May;137(5):581-93. PMID 11346336
- [Background] Girardi M, Heald PW, Wilson LD. The pathogenesis of mycosis fungoides. N Engl J Med. 2004 May 6;350(19):1978-88. doi: 10.1056/NEJMra032810. No abstract available. PMID 15128898
- [Derived] Demierre MF, Ferzli P, Miller D. Measuring HRQOL in patients with cutaneous T-cell lymphoma undergoing therapy with oral bexarotene and extracorporeal photopheresis. Arch Dermatol. 2007 May;143(5):659-61. doi: 10.1001/archderm.143.5.659. No abstract available. PMID 17515522